CLINICAL TRIAL: NCT05470816
Title: Tranexamic Acid to Reduce Delirium After Gastrointestinal Surgery: the TRIGS-D Trial (a Substudy of the TRIGS Trial)
Brief Title: Tranexamic Acid to Reduce Delirium After Gastrointestinal Surgery: the TRIGS-D Trial
Acronym: TRIGS-D
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 58/20
Record Dates: First submitted 2022-07-05; First posted 2022-07-22 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Surgical Site Infection; Dementia; Cognition
MeSH Terms: conditions — Surgical Wound Infection; Dementia | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: Multicentre, randomised, triple-blind, placebo-controlled, clinical trial (a substudy of the TRIGS trial).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: TxA blinded for the TRIGS Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic Acid (Active Comparator): 12 mg/kg, before surgical incision, and then an infusion of 3 mg/kg/h until the end of surgery.
  Interventions: Drug: Tranexamic Acid 100Mg/ml Inj Vial 10ml
- Placebo (Placebo Comparator): 12 mg/kg, before surgical incision, and then an infusion of 3 mg/kg/h until the end of surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid 100Mg/ml Inj Vial 10ml — Intervention is from the Tranexamic acid to Reduce Infection after Gastrointestinal Surgery: the TRIGS Trial. A multicentre, pragmatic, double-blind, randomised clinical trial will compare the incidence of surgical site infection and red cell transfusion requirements after IV tranexamic acid and placebo in patients undergoing gastrointestinal surgery
  Other Names: Cyklokapron
  Arms: Tranexamic Acid
Drug: Placebo — Normal saline
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
Prophylactic TxA administration in patients undergoing major gastrointestinal surgery reduces the incidence of delirium after surgery when compared with placebo. The unifying hypothesis is that systemic and neuro-inflammation lead to neuronal injury and resultant postoperative delirium.

DETAILED DESCRIPTION:
Delirium is a devastating complication of medical and perioperative care, associated with increased morbidity and mortality, dementia and impaired long-term cognition, and loss of independence. Delirium is also associated with neuronal injury placing patients at risk for long-term changes in cognition. There are no proven therapies for postoperative delirium, mainly due to the lack of adequately powered, biologically plausible trials.

There is growing evidence that tranexamic acid (TxA) may reduce inflammatory pathways in the central nervous system and protect the blood-brain barrier in trauma, and surgery.

This sub-study of the TRIGS trial (www.trigs.com.au) is evaluating the potential impact of TxA on the incidence and severity of delirium after surgery.

TRIGS-D Study Aims: In a subset of 826 patients enrolled in the TRIGS randomized trial data will be collected to identify delirium incidence and severity. The specific aims are to investigate whether TxA:

Aim 1: Reduces the incidence of postoperative delirium diagnosed with the 3D-CAM.

Aim 2: Reduces the severity of delirium diagnosed with the 3D-CAM-Severity (3D-CAM-S).

Aim 3: Modulates inflammatory (plasma cytokines, innate cell immune profile) and neurophysiological (EEG) responses in concert with any alteration in the incidence or severity of delirium.

Aim 4: Reduces longer-term impairment of quality of life and improves disability-free survival.

Primary hypothesis: Prophylactic TxA administration in patients undergoing major gastrointestinal surgery reduces the incidence of delirium after surgery when compared with placebo. The unifying hypothesis is that systemic and neuro-inflammation lead to neuronal injury and resultant postoperative delirium.

Study Design: Multicentre, randomized, triple-blind, placebo-controlled, clinical trial (a sub-study of the TRIGS trial). Patients are randomly assigned to either TxA or matched placebo. The incidence of postoperative delirium will be assessed daily using the 3D-CAM or CAM-ICU and medical record review for the first 3 days after surgery. In addition, follow up assessments will be done at 30 days and 12 months.

ELIGIBILITY:
Inclusion criteria

* Adult patients scheduled for elective gastrointestinal (oesophageal, gastric, hepatobiliary, colorectal) surgery
* with 2 or more risk factors for complications:
* age ≥70 years,
* American Society of Anesthesiologists (ASA) physical status 3 or 4,
* heart failure, diabetes,
* chronic respiratory disease,
* obesity (BMI ≥30 kg/m2),
* vascular disease,
* preoperative haemoglobin <100 g/L,
* renal impairment (se. creatinine ≥150 micromol/L), or low albumin (<30 g/L).
* Written informed consent will be obtained. Exclusion criteria
* Poor spoken and/or written language comprehension,
* laparoscopic and other minor (eg. closure of stoma) surgery,
* pre-existing infection/sepsis,
* history of spontaneous pulmonary embolism or arterial thrombosis,
* current arterial or venous thrombosis,
* familial thrombophilia (e.g. Lupus anticoagulant, protein C deficiency, factor V Leiden),
* contraindication to TxA.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 826 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-08-13 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
incidence of delirium in the first 3 days postoperatively | post surgical incision to day 3 (at anytime)obtaining information from the patient, family and staff, and thorough chart review
  3D-Confusion Assessment Method (3D-CAM) or CAM-ICU if the Used to measure delirium. Assessments will be conducted twice daily A classification of delirium will be made if both features 1 and 2 are present

SECONDARY OUTCOMES:
Delirium severity | post surgical incision to day 3 (inclusive)
  3D-CAM-S
Quality of Life Intergroup differences | 12 months post surgical incision
  using the Short form survey 12 - Quality of Life Intergroup differences in long-term (12 month) in perioperative cognitive decline
Disability | 12 months post surgical incision
  World Health Organization disability assessment schedule. Intergroup differences in long-term (12 month) in perioperative cognitive decline
perioperative neurocognitive disorders (NCDs) | 12 months post surgical incision
  NCD will be defined as any of: (i) subjective complaint, (ii) a 4-point reduction in TICS-B, (iii) SF or VF, and (iv) functional deficit defined as a reduction in WHODAS score of 5% or more from baseline (before surgery).
Days at home up to 30 days after surgery (DAH30) | 30 days post surgical incision post surgical incision
  DAH30 is patient-centred and reflects the patient's primary aim of a healthy recovery, reduced hospital costs and serious complications, and avoiding re-admission (often due to postoperative delirium).
cytokine levels | preoperative, postoperative day 1 and 3 post surgical incision
  Blood tests measured in 92 key inflammatory/immune markers using technology
neuronal injury biomarker | preoperative, postoperative day 1 and 3 post surgical incision
  used to evaluate temporal changes in the innate cellular immune and inflammatory profile, and for changes in fibrinolysis

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Myles, DSci, Study Chair — Monash University
Locations (1):
- Alfred Health, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Following written request and review by the steering committee
Supporting Information: Study Protocol, SAP
Time Frame: Following analysis for the publication
Access Criteria: Written request